CLINICAL TRIAL: NCT01638286
Title: Study to Evaluate a Pharmacokinetic Drug Interaction Between Eperisone Hydrochloride and Aceclofenac in Healthy Male Subjects
Status: Completed | Type: Observational
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: HM-EPAC-101
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Acute Low Back Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Eperisone
- Aceclofenac
- Eperisone hydrochloride, Aceclofenac

SUMMARY:
A randomized, open label, single-dose, 6-sequence, 3-period, crossover study to evaluate a pharmacokinetic drug interaction between eperisone hydrochloride and aceclofenac in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI : 20.0 - 28.0 kg/m2 willingness to sign the written informed consent form(ICF)

Exclusion Criteria:

* Evidence of clinically relevant pathology within 30 days prior to drug administration History of relevant drug and/or food allergies

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Acute low back pain
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)